CLINICAL TRIAL: NCT05458037
Title: A Randomized Controlled Trial of Pain Perception With Fast and Slow Tenaculum Application to the Uterine Cervix
Brief Title: RCT of Pain Perception With Fast and Slow Tenaculum Application
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1609832
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Pain, Acute; Pain, Procedural
MeSH Terms: conditions — Acute Pain; Pain, Procedural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast tenaculum application (Experimental)
  Interventions: Procedure: Speed of tenaculum application
- Slow tenaculum application (Experimental)
  Interventions: Procedure: Speed of tenaculum application

INTERVENTIONS:
Procedure: Speed of tenaculum application — Fast or slow closure of the tenaculum for application to the uterine cervix

SUMMARY:
This project will be a randomized controlled trial (RCT) measuring pain perception with two different tenaculum placement techniques on the uterine cervix. A tenaculum is an instrument used to hold the cervix (the opening to the uterus or womb) in place. The trial will measure pain perception with a Visual Analog Scale (VAS) from 0 to 100 mm for two different tenaculum placement techniques, fast and slow closure on the uterine cervix. The main objective of this study is to determine if there is a difference in pain perception with fast compared to slow tenaculum placement techniques on the uterine cervix. We hypothesize that the slow technique will be perceived as less painful for subjects as measured on a 0 mm to 100 mm Visual Analog Scale (VAS). Subsidiary objectives include describing overall pain levels during the procedure.

DETAILED DESCRIPTION:
In order to detect a 15 mm difference on the VAS with two-sided 5% alpha and 80% power and a standard deviation of 33 mm (based on prior studies), a total of 71 subjects per group are required. We aim to recruit 75 subjects per arm in order to account for possible drop out.

ELIGIBILITY:
Inclusion Criteria:

1. plans for IUD insertion or endometrial biopsy;
2. 18 to 49 years of age;
3. not taken analgesics or anxiolytics in the previous 24 hours;
4. the ability and are willing to give informed consent.

Exclusion Criteria:

1. Do not speak English unless interpreter present;
2. Taken any narcotic or opiate medication in the last 24 hours.
3. Taken any recreational or illegal drugs in the last 24 hours, such as marijuana, heroin, cocaine, crack, or methamphetamines.
4. Taken any anti-anxiety medication or drug in the last 24 hours.
5. Taken any NSAIDS or Tylenol in the last 12 hours.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain perception with tenaculum application | during procedure
  Pain scores will be determined using the Visual Analog Scale (VAS) from 0 to 100 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Allen, MD, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RH, Micks E, Edelman A. Pain relief for obstetric and gynecologic ambulatory procedures. Obstet Gynecol Clin North Am. 2013 Dec;40(4):625-45. doi: 10.1016/j.ogc.2013.08.005. PMID 24286993
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Doty N, MacIsaac L. Effect of an atraumatic vulsellum versus a single-tooth tenaculum on pain perception during intrauterine device insertion: a randomized controlled trial. Contraception. 2015 Dec;92(6):567-71. doi: 10.1016/j.contraception.2015.05.009. Epub 2015 May 22. PMID 26007292
- [Background] Ireland LD, Allen RH. Pain Management for Gynecologic Procedures in the Office. Obstet Gynecol Surv. 2016 Feb;71(2):89-98. doi: 10.1097/OGX.0000000000000272. PMID 26894801
- [Background] Lambert T, Truong T, Gray B. Pain perception with cervical tenaculum placement during intrauterine device insertion: a randomised controlled trial. BMJ Sex Reprod Health. 2020 Apr;46(2):126-131. doi: 10.1136/bmjsrh-2019-200376. Epub 2019 Oct 30. PMID 31666302